CLINICAL TRIAL: NCT06105411
Title: Siderophore-labelled Positron Emission Tomography for Correlating Invasive Fungal InfeCtions
Acronym: SPECIFIC
Status: Recruiting | Type: Observational
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Other Study IDs: SPECIFIC
Record Dates: First submitted 2023-10-12; First posted 2023-10-27 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Invasive Fungal Infections
Keywords: Invasive Fungal Infections; Siderophore; PET; Siderophore-labelled Position Emission tomography; 68Ga-labelled TAFC PET/CT scan; Aspergillus spp.
MeSH Terms: conditions — Invasive Fungal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: 68Ga-labelled TAFC PET/CT scan — 68Ga-labelled TAFC PET/CT scan (whole body)

SUMMARY:
This trial will demonstrate localised uptake of a radiolabelled fungal component (siderophore) in areas of known specific invasive fungal (Aspergillus) infection.

DETAILED DESCRIPTION:
This open label, single centre, proof of concept pilot imaging trial will evaluate technique for the diagnosis of invasive Aspergillus infection. It aims to demonstrate uptake of the gallium-siderophore tracer at sites of known proven/probable invasive aspergillus app infection. It will also assess the safety and tolerability of this technique.

10 patients within 2 weeks of proven or probable invasive fungal infection (IFI) diagnosis will be recruited to this study over a period of 12-24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has provided written informed consent
2. Aged 18 years or older at written informed consent
3. Within 2 weeks of proven or probable or possible invasive fungal infection (IFI) diagnosis as per EORTC criteria
4. Imaging consistent with invasive pulmonary aspergillosis on CT or FDG-PET/CT with lesions at least 8mm in diameter
5. Patient is willing and able to comply with the protocol for the duration of the study including scheduled visits such as follow up

Exclusion Criteria:

1. Women who are pregnant or lactating.
2. Iron infusion within one week prior to scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older at written informed consent who have proven or probable invasive fungal infection (IFI) diagnosis with imaging consistent with invasive pulmonary aspergillosis on CT or FDG-PET/CT with lesions at least 8mm in diameter. They are also willing and able to comply with the protocol for the duration of the study including scheduled visits such as follow up.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Uptake of radiolabelled siderophore (68Ga-TAFC) in patients with proven/probable invasive Aspergillosis | At 60 minutes
  The maximum standardized uptake value (SUVmax) is widely used for measuring the uptake of FDG by malignant tissue.

SECONDARY OUTCOMES:
Physiologic bio distribution | Evaluated up to 3 hours following injection of radiotracer
  SUVmax in mediastinal blood pool, and any organs with uptake including liver, spleen and marrow
Safety of 68Ga-TAFC-PET/CT | Evaluated within 24 hours of scan
  Adverse events defined by CTCAE v5
Findings compared to CT and/or 18F-FDG PET/CT | At 60 minutes
  Descriptive comparison of the siderophore PET to standard of care imaging - looking at areas of uptake and if this corresponds to areas of presumed infection on SOC PET or CT

CONTACTS AND LOCATIONS:
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia